CLINICAL TRIAL: NCT03758729
Title: Phase II Study of Nivolumab in Combination With Radiation Therapy as Definitive Treatment for Patients With Locally Advanced, Unresectable Head and Neck Mucosal Melanoma.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Internal Issues
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD, PhD, Division of Hematology-oncology, Department of medicine, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-04-093
Record Dates: First submitted 2018-11-28; First posted 2018-11-29 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab 3mg/kg + NS 100mL MIV over 1hr every 2 weeks
  Interventions: Drug: Nivolumab; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Nivolumab — Nivolumab 3mg/kg + NS 100mL MIV over 1hr every 2 weeks
Radiation: Radiation Therapy — Radiation Therapy

SUMMARY:
This is a Phase 2, single center study to evaluate the efficacy, safety of nivolumab in combination with radiation therapy in patients with mucosal melanoma of the head and neck (MMHN). Target Accrual and Study duration We will accrue up to 26 patients. It is estimated to take up to 2 years. The sample size is calculated by use of SWOG CRAB (Cancer Research And Biostatistics) to control the type I error at 5 % for null hypothesis that the true response rate was 25 % or below and to have 80 % of power if the true response rate was 50 % or higher. Although the target number of evaluable patients is 23, we planned to recruit 10% more than the target number of patients considering dropout, total 26.

DETAILED DESCRIPTION:
This is a phase II, single-arm, single-center study to evaluate the response rate, efficacy and safety of nivolumab in combination with radiation therapy in subjects with of locally advanced, unresectable head and neck mucosal melanoma.

A cycle is defined as 14 days. The nivolumab dose will be fixed at the recommended phase II dose of 3mg/kg as a 60-minute IV infusion every two weeks. Patients will continue on nivolumab up to 8 weeks, until disease progression, unacceptable toxicity, investigator's decision to remove patient from the study, patient refusal to continue, or alternative treatment.

Concurrent radiotherapy of 70Gy for 6-7 weeks will be initiated on the same day of first nivolumab dose of cycle 1.

The combination of 70 Gy radiotherapy for 6-7 weeks begins on the day of initial administration of nivolumab, radiation therapy dose and treatment schedule 2.0, based on NCFC practice.

Nivolumab is administered every two weeks in in combination with radiation therapy and has elapsed since 8 weeks (after 4 cycles) The administration of clinical trials in is terminated but nivolumabs is sustainable at the discretion of investigator. (This is carried out independently of the clinical trial) The response rate of radiation therapy is assessed by performing a tumor assessment every two months up to the end of radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years
* Histologically or cytologically confirmed mucosal melanoma of head and neck
* Locally advanced and unresectable
* No previous chemotherapy for purpose of palliation
* ECOG performance status of 0~2
* Measurable lesion per RECIST 1.1 criteria
* Be willing to provide fresh tissue for biomarker analysis, and, based on the adequacy of the tissue sample quality for assessment of biomarker status. Repeat samples may be required if adequate tissue is not provided. Newly obtained endoscopic biopsy specimens are preferred to archived samples and formalin-fixed, paraffin-embedded (FFPE) block specimens are preferred to slides.
* Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen.
* Collection of an archived tissue sample will also be requested (where available) to support evaluation of the clinical utility of biomarker assessment in newly obtained vs. archived tissue samples; however, a subject will not be precluded from participating in the study if an archived tissue sample is not available for collection or is otherwise insufficient for analysis.
* Adequate marrow, hepatic, renal and cardiac functions:

Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN), or AST and ALT ≤ 5 x ULN if liver function abnormalities are due to underlying malignancy Total serum bilirubin ≤ 1.5 x ULN Absolute neutrophil count (ANC) ≥ 1,500/uL Platelets ≥ 100,000/uL Hemoglobin ≥ 8.0 g/dL Serum creatinine OR Measured or calculateda creatinine clearance (GFR can also be used in place of creatinine or CrCl) Serum creatinine ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN

* Creatinine clearance should be calculated per institutional standard.

  * Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
  * Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 8.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
  * Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
  * provision of a signed written informed consent

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Active or history of autoimmune disease or immune deficiency, including MG, myositis, hepatitis, SLE, RA, IBD or GBS)
* Severe co-morbid illness and/or active infections
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has a known history of active TB (Bacillus Tuberculosis)
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Pregnant or lactating women
* History of documented congestive heart failure; angina pectoris requiring medication; evidence of tranasmural myocardial infarction on ECG; poorly controlled hypertension; clinically significant valvular heart disease; or high risk of uncontrollable arrhythmia
* Active CNS metastases not controllable with radiotherapy or corticosteroids (however, CNS metastases (except for leptomeningeal seeding) are allowed if controlled by gamma knife surgery or surgery or radiotherapy or steroid)
* Must not have undergone a major surgical procedure < 4 weeks or radiotherapy <2 weeks prior to D1 of treatment
* Administration of a live, attenuated vaccine within 4 weeks before study treatment
* Treatment with systemic immunosuppressive medication (including prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, anti-tumor necrosis factor agents) within 2 weeks prior to D1 of treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Response rate | 2 years
  RR, as determied by irRECIST criteria, is defined as the proportion of all subjects whose best overall response (BOR) is either a CR or PR. BOR is determined by the best response designation recorded between the date of treatment initiation and the date of first objectively documented progression or the date of subsequent anti-cancer therapy, whichever is the first. For subjects without documented progression or subsequent anti-cancer therapy, all available repsonse designations will contribute to the BOR determination.